CLINICAL TRIAL: NCT06409585
Title: Cardiomyopathies and Heart Muscle Diseases: Cardiac Imaging in the Evaluation of Myocardial Fibrosis Transition
Acronym: CHIEFTain
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 307358
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Hypertrophic Cardiomyopathy; Cardiac Sarcoidosis; Hypertensive Heart Disease; Tako Tsubo Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy 1; Myocarditis
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Takotsubo Cardiomyopathy; Arrhythmogenic Right Ventricular Dysplasia, Familial, 1; Myocarditis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Heart failure with preserved ejection fraction: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI
- Hypertrophic cardiomyopathy and Hypertensive heart disease: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI
- Cardiac Sarcoidosis: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI
- Arrhythmogenic cardiomyopathy: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI
- Myocarditis: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI
- Takotsubo cardiomyopathy: Participants will undergo baseline echocardiography and hybrid cardiac PET-MR with 200MBq of 68Ga-FAPI or 18F-AlF-FAPI. A follow-up echocardiogram and cardiac MRI will be undertaken a year later.
  Interventions: Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR; Diagnostic Test: Echocardiogram; Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI or 18F-AlF-FAPI cardiac PET-MR — 200MBq of the above named radiotracer will be administered for PET-MR
Diagnostic Test: Echocardiogram — Echocardiogram at baseline and 1 year follow-up
Diagnostic Test: Cardiac MRI — Cardiac MRI at 1 year

SUMMARY:
Heart scarring, also known as fibrosis, plays a major role in a lot of heart muscle abnormalities. These abnormalities of the heart muscle can lead to major issues such as symptoms of heart failure, dangerous heart rhythm disturbances and even death. However, a lot of these conditions are still not fully understood and treatment options are limited. We here aim to use a new radioactive dye called 68Ga-FAPI to identify patterns and the activity of heart muscle scarring. This radioactive dye is being used in humans particularly in identifying and monitoring cancers and has shown promise in identifying scarring in the heart as well. This will help us not only understand the underlying disease process and risk stratify these patients but also potentially help us develop new targeted therapies that can affect heart muscle scarring. Participants will undergo a baseline MRI scan using this new dye and a plain MRI scan will repeated 12-18 months after to see if there are any changes in the process.

ELIGIBILITY:
Inclusion Criteria:

HFpEF cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Patients with symptomatic heart failure with preserved ejection fraction as defined by the presence of heart failure symptoms (dyspnoea, reduced exercise tolerance, fatigue), signs (elevated jugular venous pressure, pulmonary crackles, peripheral oedema) as well as echocardiographic features (preserved left ventricular systolic function (>50%) and reduced diastolic function with septal e' <7cm/s or lateral e' <10cm/s).

Hypertrophic cardiomyopathy cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Established diagnosis of hypertrophic cardiomyopathy: left ventricular wall thickness >15mm by any imaging modality without a loading condition to explain the hypertrophy OR
* Left ventricular wall thickness of >13 mm by any imaging modality in the presence of a genetic or non-genetic component, supported by other features including family history, non-cardiac symptoms, ECG changes and laboratory tests.

Hypertensive heart disease cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Diagnosis of essential hypertension for at least 1 year with evidence of left ventricular hypertrophy on echocardiography (left ventricular mass index >98 g/m2 and relative wall thickness >0.42)

Arrhythmogenic cardiomyopathy

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Diagnosis of arrhythmogenic right ventricular cardiomyopathy based on the International Task Force 2010 criteria

Myocarditis cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Diagnosis of myocarditis in the past month defined with the following features

  * Chest pain
  * Evidence of pericarditis (pericardial rub, ST- segment elevation or pericardial effusion)
  * Elevated serum troponin
  * Unobstructed coronary arteries on coronary angiogram OR
  * Cardiac magnetic resonance imaging evidence of myocarditis (subepicardial or mid-wall late gadolinium enhancement

Takotsubo cardiomyopathy cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Diagnosis of takotsubo cardiomyopathy in the past month as defined by European Society of Cardiology guidelines 2018

Cardiac sarcoidosis cohort

* Male or female between 30 to 90 years old
* Provision of informed consent prior to any study specific procedures
* Diagnosis of cardiac sarcoidosis for at least 1 year based on expert consensus opinion with

  * Histological diagnosis from a myocardial biopsy OR
  * Histological diagnosis of extra-cardiac sarcoid AND

One or more of following is present

* Steroid +/- immunosuppressant responsive cardiomyopathy or heart block
* Unexplained reduced LVEF (<40%)
* Unexplained sustained (spontaneous or induced) VT
* Mobitz type II 2nd degree heart block or 3rd degree heart block
* Patchy uptake on dedicated cardiac PET (in a pattern consistent with CS)
* Late Gadolinium Enhancement on CMR (in a pattern consistent with CS)
* Positive gallium uptake (in a pattern consistent with CS) AND
* Other causes for the cardiac manifestation(s) have been reasonably excluded

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* History of claustrophobia or inability to tolerate supine position for the PET/MR or PET/CT scans.
* Impaired renal function with eGFR of <30 mL/min/1.73 m2.
* Women who are pregnant or breastfeeding.
* Iodine or gadolinium contrast allergy
* Contra-indication to CT scanning

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As highlighted in the inclusion criteria above
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Standardised uptake values | 1-2 years
Target-to-background ratio | 1-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other research groups